CLINICAL TRIAL: NCT03266692
Title: A Phase 1 Study of ACTR087, an Autologous T Cell Product, in Combination With SEA-BCMA, a Monoclonal Antibody, in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of ACTR087 in Combination With SEA-BCMA in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Cogent Biosciences, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATTCK-17-01
Record Dates: First submitted 2017-08-22; First posted 2017-08-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Refractory Multiple Myeloma
Keywords: BCMA; SEA-BCMA; B Cell Maturation Antigen; ACTR; ACTR087; T cell; T cell product; relapsed; refractory; multiple myeloma; adoptive T cells; autologous; gene therapy; cell therapy
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACTR087 in combination with SEA-BCMA (Experimental)
  Interventions: Biological: ACTR087; Biological: SEA-BCMA

INTERVENTIONS:
Biological: ACTR087 — Autologous T cell product
Biological: SEA-BCMA — B-cell maturation antigen (BCMA)-directed antibody

SUMMARY:
This is a phase 1, multi-center, single-arm, open-label study evaluating the safety, tolerability, and anti-myeloma activity of ACTR087 (an autologous T cell product) in combination with SEA-BCMA (a monoclonal antibody) in subjects with relapsed or refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures
* Histologically- or cytologically-confirmed relapsed or refractory multiple myeloma (MM) with measurable disease
* Must have received at least 3 prior lines of therapy to include treatment with a proteasome inhibitor (eg, bortezomib, carfilzomib, or ixazomib) and an immunomodulatory agent (eg, lenalidomide, pomalidomide) unless double-refractory to both; and a hematopoietic stem cell transplant (HSCT), for those subjects considered HSCT-eligible.
* Quantitative serum IgG levels for subjects with IgG MM must not exceed the institutional upper limit of normal (ULN)
* ECOG 0 or 1
* Life expectancy of at least 6 months
* Absolute neutrophil (ANC) count greater than 1000/ µL
* Platelet count greater than 50,000/µL
* Estimated GFR >30mL/min/1.73m2

Exclusion Criteria:

* Known active central nervous system (CNS) involvement by MM
* Systemic rheumatic or autoimmune diseases or acute or chronic infections
* Uncontrolled thromboembolic events or recent severe hemorrhage
* Subjects who are currently using more than 5mg/day of prednisone (or an equivalent glucocorticoid exceeding physiologic replacement levels)
* Prior treatment as follows:

  * T cell-directed antibody therapy (eg. Alemtuzumab, anti-thymocyte globulin) within 6 months of enrollment
  * Any prior myeloma-directed therapy including cytotoxic chemotherapy, biologic therapy, or radiotherapy within 2 weeks of enrollment
  * Any mAb or other protein therapeutic containing Fc-domains within 4 weeks of enrollment
  * Experimental agents within 3 half-lives prior to enrollment, unless progression is documented on therapy
  * Prior BCMA-directed investigational agents at any time
  * Prior cell or gene therapy, excluding transfers of genetically unmodified autologous cells (eg. Hematopoietic stem cell transplantation), at any time; or prior allogeneic HSCT at any time
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ACTR087 in combination with SEA-BCMA | 28 days
  Composite outcome measure assessed by committee review of dose limiting toxicities (DLTs), incidence and severity of AEs and clinically significant abnormalities of laboratory values
Determination of recommended Phase 2 dosing regimen | 52 weeks
  Review of DLTs, Maximum tolerated contour (MTC), incidence and severity of AEs and clinically significant abnormalities of laboratory values

SECONDARY OUTCOMES:
Safety of SEA-BCMA as measured by incidence of Treatment Emergent Adverse Events (TEAEs) | 21 days
  Review of all TEAEs, including incidence and severity of AEs, DLTs and clinically significant abnormalities of laboratory values
Anti-myeloma activity as measured by overall response rate (per IMWG response criteria) | 52 weeks
Anti-myeloma activity as measured by duration of response | 52 weeks
Anti-myeloma activity as measured by progression-free survival | 52 weeks
Anti-myeloma activity as measured by overall survival | 52 weeks
Assessment of persistence of ACTR087 as measured by flow cytometry and qPCR | 52 weeks
Assessment of ACTR087 phenotype and function as measured by flow cytometry | 52 weeks
Assessment of induction of inflammatory markers and cytokines/chemokines after ACTR087 administration | 52 weeks
  Levels of inflammatory markers, cytokines/chemokines
SEA-BCMA PK | 52 weeks
  SEA-BCMA plasma concentration
Assessment of anti-drug antibodies (ADA) after SEA-BCMA administration | 52 weeks
  Incidence of ADAs to SEA-BCMA

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sachs, MD, Study Director — Cogent Biosciences, Inc.
Locations (7):
- United States (7):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Baylor Scott & White, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin